CLINICAL TRIAL: NCT05096520
Title: The Efficiency of Radiofrequency Ablation Therapy Applied to the Intermedius Genicular Nerve in the Treatment of Patients With Chondromalacia Patella
Brief Title: Intermedius Genicular Nerve in the Treatment of Patients With Chondromalacia Patella
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Physical Medicine and Rehabilitation Specialist, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19
Record Dates: First submitted 2021-09-20; First posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Chondromalacia Patellae
Keywords: radiofrequency neurotomy; knee pain; ultrasound
MeSH Terms: conditions — Chondromalacia Patellae | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- radiofrequency group (Active Comparator): the radiofrequency needle will be advanced percutaneously towards the intermedius genicular nerve on the periosteum of the distal femoral shaft region until bone contact is achieved. In addition to imaging the nerve with ultrasound, sensory stimulation at 50 Hz frequency will be applied with a threshold value less than 0.6 V in order to determine its position more accurately. In order to prevent the inactivation of the motor nerves, the relevant nerve will be tested for the absence of fasciculation in the region of the lower extremity compatible with the application with the stimulation with a frequency of 2.0 V and 2 Hz. Before the activation of the radiofrequency generator, an injection of 1 ml of 2% lidocaine will be made, then the radiofrequency electrode will be added to the needle and the temperature level at the tip of the electrode will be increased to 80 degrees for 2 minutes, the procedure will be performed for each genicular nerve.
  Interventions: Procedure: radiofrequency; Drug: 2% lidocaine
- control group (Active Comparator): The intermedius genicular nerve will be found under US guidance and the genicular nerve will be blocked by injecting 1 ml of 2% lidocaine.
  Interventions: Procedure: control; Drug: 2% lidocaine

INTERVENTIONS:
Procedure: radiofrequency — the radiofrequency needle will be advanced percutaneously towards the intermedius genicular nerve on the periosteum of the distal femoral shaft region until bone contact is achieved. In addition to imaging the nerve with ultrasound, sensory stimulation at 50 Hz frequency will be applied with a threshold value less than 0.6 V in order to determine its position more accurately. In order to prevent the inactivation of the motor nerves, the relevant nerve will be tested for the absence of fasciculation in the region of the lower extremity compatible with the application with the stimulation with a frequency of 2.0 V and 2 Hz. Before the activation of the Baylis brand radiofrequency generator, an injection of 1 ml of 2% lidocaine will be made, then the radiofrequency electrode will be added to the needle and the temperature level at the tip of the electrode will be increased to 80 degrees for 2 minutes, the procedure will be performed for each genicular nerve.
  Arms: radiofrequency group
Procedure: control — The intermedius genicular nerve will be found under US guidance and the genicular nerve will be blocked by injecting 1 ml of 2% lidocaine.
  Arms: control group
Drug: 2% lidocaine — 2% lidocaine

SUMMARY:
Radiofrequency application is a treatment method that temporarily prevents the transmission of pain in the nerve where the application is made through the heat emitted by radio waves.Partial inhibition of the functions of the nerves carrying the joint pain sensation with this method is the basis of the treatment.The intermedius genicular nerve carries the sensation of subpatellar pain due to chondromalacia.In this study,investigators aim is to investigate the effect of radiofrequency neurotomy applied to the intermedius genicular nerve, which receives the sensation of the patella, on pain and knee function in patients with a diagnosis of chondromalacia patella who have anterior knee pain that does not resolve despite conservative treatment, under the guidance of ultrasonography.

DETAILED DESCRIPTION:
The study was designed as prospective, randomized, controlled trial. 46 people who met the inclusion criteria were randomized into two groups of 23 people. The first group will be designated as Nerve blockage group and nerve blocking program will be applied to these patients. Patients in the second group will be designated as the Radiofrequency group and radiofrequency ablation after the blockade program will be applied in accordance with the radiofrequency ablation protocol.Participants were evaluated with Visual Analogue Scale (VAS), Patello Femoral Pain Severity Scale (PFPSS), Kuala's Patellofemoral Scoring System (KPSS).

ELIGIBILITY:
Inclusion Criteria:

* Male/female aged >18 years
* Diagnosis of chondromalacia patella after physical examination and MR imaging
* Those whose symptoms persist for >3 months
* Participating in the study voluntarily

Exclusion Criteria:

* Pregnant patients
* History of previous knee surgery
* To have received physical therapy from the knee area in the last 6 months
* Previous RF treatment or any therapeutic injection of the knee such as steroid, hyaluronic acid within 3 months
* Those with pain radiating from the waist or hip
* Patients with neuropathic pain
* History of tumor, infectious, psychiatric disease, bleeding diathesis
* History of knee trauma in the last 6 months
* Those with systemic diseases such as hepatitis, coagulopathy
* Patients with BMI >40
* Finding a leg length difference

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-07-15 (Estimated)

PRIMARY OUTCOMES:
Knee Pain Severity of pain was assessed using the standard 10 cm VAS with 0 meant "no pain" at one end, and 10 meant "unbearable pain" at the other end initial, 4th week 7th week 24th week pain change | Change from Baseline , 4th week 12th week
  Severity of pain was assessed using the standard 10 cm VAS with 0 meant "no pain" at one end, and 10 meant
  "unbearable pain" at the other end

SECONDARY OUTCOMES:
Patello Femoral Pain Intensity Scale | Change from Baseline, 4th week 12th week
  Patello Femoral Pain Intensity Scale to evaluate patients' pain in climbing / descending stairs, squatting, walking, jogging, sprinting, sports, sitting for 20 minutes with knees flexed at 90 °, standing on the knee, resting and resting after an activityStair climbing / descending, crouching, walking, jogging, sprinting, sports, sitting for 20 minutes with knees flexed at 90 °, standing on the knee, resting and resting after an activity, travel 10 cm as standard 0 "no pain" at one end, 10 At the other end it was rated as "excruciating pain" with a total score of 100.

OTHER OUTCOMES:
Kuala Patellofemoral Scoring System | Change from Baseline, 4th week 12th week
  Kuala Patellofemoral Scoring System was used to determine the functional levels of the patients. Participants were evaluated over a minimum of 0 and a maximum of 100 points

CONTACTS AND LOCATIONS:
Overall Officials: Serdar KESİKBURUN, MD, Study Director — SBU,Gaziler Physical Medicine and Rehabilitation Education and Research Hospital; Burak BAYIR, MD, Principal Investigator — SBU,Gaziler Physical Medicine and Rehabilitation Education and Research Hospital; Özlem KÖROĞLU, MD, Principal Investigator — SBU,Gaziler Physical Medicine and Rehabilitation Education and Research Hospital; Esra ÇELİK KARBANCIOĞLU, MD, Principal Investigator — SBU,Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Locations (1):
- Gaziler Physical Medicine and Rehabilitation Education and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No